CLINICAL TRIAL: NCT01508676
Title: Effects of Pennsaid on Clinical Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jianren Mao, MD, PhD, Vice Chair Research, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 2011p000897
Record Dates: First submitted 2012-01-04; First posted 2012-01-12 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Neuralgia; Postherpetic Neuralgia; Reflex Sympathetic Dystrophy; Complex Regional Pain Syndrome (CRPS)
Keywords: neuropathic pain; postherpetic neuralgia; complex regional pain syndrome; reflex sympathetic dystrophy
MeSH Terms: conditions — Neuralgia; Neuralgia, Postherpetic; Reflex Sympathetic Dystrophy; Complex Regional Pain Syndromes | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pennsaid Phase I (Active Comparator): Pennsaid (20-40 drops; 2-4 times daily) Upon completion of the first phase, subjects in each arm will be crossed over (i.e., from placebo to Pennsaid and vise versa). Pennsaid or placebo lotion will be packed in a container with identical appearance before being dispensed to study subjects.
  Interventions: Drug: Pennsaid
- Placebo Phase I (Placebo Comparator): Study subject will topically apply placebo lotion (20-40 drops) 2-4 times daily to the painful area for the next two weeks. The dose titration will be based on the size of painful area (approximately 10 drops for every 4 square inches). Subjects will be asked to fill in a daily pain diary and report any side effects to the research center. A phone number and a beeper number will be provided to subjects.
  Interventions: Drug: Placebo (2.3% DMSO solution)

INTERVENTIONS:
Drug: Pennsaid
  Other Names: Pennsaid topical 1.5% diclofenac; a non-steroid anti-inflammatory drug
  Arms: Pennsaid Phase I
Drug: Placebo (2.3% DMSO solution)
  Other Names: Placebo (2.3% DMSO solution; 20-40 drops; 2-4 times daily).
  Arms: Placebo Phase I

SUMMARY:
The purpose of this study is to see if the drug Pennsaid (Diclofenac) can help reduce pain felt by people with chronic nerve pain. The drug will be used 2-4 times each day for 2 weeks.

The U.S. Food and Drug Administration (FDA) has approved Pennsaid to treat osteoarthritis (bone pain), but the FDA has not approved Pennsaid to treat neuropathic (nerve) pain.

The research study will compare Pennsaid to placebo.

DETAILED DESCRIPTION:
The research study will compare Pennsaid to placebo. The placebo looks like Pennsaid, but it doesn't contain any Pennsaid. The investigators use placebos in research to see if the results are due to the study drug or to other reasons. At some time during the study the investigators will give the patient Pennsaid. At another time, the investigators will give the patient placebo. The investigators are using Quantitative Sensory Testing (QST), which is temperature testing before and after using the study drug to see if Pennsaid is helpful in reducing people's nerve pain.

In this test, a small metal plate, about the size of a matchbox, is put on the area where the patient has pain. The plate is connected to a computer that can warm or cool the plate. The patient will use a computer mouse button to tell us when the plate feels warm. The QST machine is approved by the Food and Drug Administration (FDA). It is often used by nerve doctors to see if a person has neuropathy (pain caused by damage to a nerve).

ELIGIBILITY:
Inclusion Criteria:

1. Subject will be between 18 and 80 years of age.
2. Subject has not been on Pennsaid or other topical non-steroid anti-inflammatory drugs for at least one month.
3. Subject agrees to make no change in his/her current pain medications during the entire study period. This requirement will ensure that valid comparisons of primary and secondary measures can be made before and after the study.
4. Subject has a VAS pain score of 4 or above at the beginning of the study.
5. Subject has had a neuropathic pain condition such as those listed above for at least three months. This requirement is to avoid clinical uncertainty from an unstable pain condition and to minimize the study variation.
6. Female subjects of childbearing age must have a negative urine pregnancy test at the initial visit.

Exclusion Criteria:

1. Subject has documented severe liver or renal disease that will affect the elimination of Pennsaid or is subject to the adverse effect of Pennsaid on these organs. (Renal dysfunction is defined as eGFR < 60. Hepatic dysfunction is defined as LFTs ≥ 3X ULN.)
2. Subject has pending litigation related to the neuropathic pain condition.
3. Subject has active skin lesion or open wound at the site of Pennsaid application (e.g., active shingles with skin lesions).
4. Subject is pregnant or lactating.
5. Subject has scar tissue or sensory deficit at the site of QST.
6. Subject is allergic to diclofenac or has cross-sensitivity to other non-steroid anti-inflammatory drugs.
7. Subject has a positive urine (illicit) drug test.
8. Subjects who experience asthma, urticaria or an allergic type reaction when taking aspirin or NSAIDs.
9. Subjects undergoing coronary artery bypass surgery.
10. Subject with a known history of cardiovascular disease, ulcer, gastrointestinal bleed or impaired renal function.
11. Subjects currently using NSAIDS.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianren Mao, M.D., Ph.D., Principal Investigator — DACCPM
Locations (1):
- MGH Center for Translational Pain Research, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pennsaid Phase I, Placebo Phase II: Phase I: 2 weeks applying Pennsaid lotion (20-40 drops; 2-4 times daily).
  Washout: 1 week, applying nothing.
  Phase II: 2 weeks applying Placebo lotion (20-40 drops; 2-4 times daily).
- Placebo Phase I, Pennsaid Phase II: Phase I: 2 weeks applying Placebo lotion (20-40 drops; 2-4 times daily).
  Washout: 1 week, applying nothing.
  Phase II: 2 weeks applying Pennsaid lotion (20-40 drops; 2-4 times daily).
Period: Phase I (2 Weeks)
Arm/Group | Pennsaid Phase I, Placebo Phase II | Placebo Phase I, Pennsaid Phase II
Started | 18 | 17
Completed | 16 | 14
Not Completed | 2 | 3
Not completed — Medication Exclusion | 1 | 1
Not completed — Wrong Pain Type | 1 | 0
Not completed — Positive Drug Screen | 0 | 2
Period: Washout Period (1 Week)
Arm/Group | Pennsaid Phase I, Placebo Phase II | Placebo Phase I, Pennsaid Phase II
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0
Period: Phase II (2 Weeks)
Arm/Group | Pennsaid Phase I, Placebo Phase II | Placebo Phase I, Pennsaid Phase II
Started | 16 | 14
Completed | 15 | 13
Not Completed | 1 | 1
Not completed — Skin Sensitivity | 0 | 1
Not completed — Medication Exclusion | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pennsaid Phase I: Pennsaid (20-40 drops; 2-4 times daily). Upon completion of the first phase, subjects in each arm will be crossed over (i.e., from placebo to Pennsaid and vise versa). Pennsaid or placebo lotion will be packed in a container with identical appearance before being dispensed to study subjects.
- Placebo Phase I: Placebo lotion (20-40 drops; 2-4 times daily). Upon completion of the first phase, subjects in each arm will be crossed over (i.e., from placebo to Pennsaid and vise versa). Pennsaid or placebo lotion will be packed in a container with identical appearance before being dispensed to study subjects.
- Total: Total of all reporting groups
Arm/Group | Pennsaid Phase I | Placebo Phase I | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 15 | 32
  >=65 years | 1 | 2 | 3
Gender [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: VAS After Treatment
Description: Subjects rated their pain using the Visual Analog Scale after a 2 week phase of using pennsaid lotion and after a 2 week phase of using placebo lotion.
  The Visual Analog Scale is subject reported on a scale of 0-10 with 0 being no pain, and 10 being the worst pain they can imagine. Results reported are an average of reported VAS scores for the 28 subjects who completed both phase I and phase II of the study.
Time Frame: 2 weeks.
Population: Only subjects who completed both phases of the crossover study were considered for data analysis.
Measure: Mean (Standard Deviation); unit: Visual Analog Scale
Groups:
- Pennsaid; Placebo: All subjects who recieved Pennsaid lotion in either Phase I or II were considered.
Arm/Group | Pennsaid | Placebo
Number analyzed (Participants) | 28 | 28
Visual Analog Scale | 4.9 (1.9) | 5.6 (2.1)
Statistical Analysis 1: Comparison: Pennsaid vs Placebo; Test type: Superiority or Other; p = .04, t-test, 2 sided

2. Secondary Outcome: Clinical Neuropathic Pain Features- Burning After Treatment
Description: Subjects rated their "burning pain" using the Visual Analog Scale after a 2 week phase of using pennsaid lotion and after a 2 week phase of using placebo lotion.
  The Visual Analog Scale is subject reported on a scale of 0-10 with 0 being no pain, and 10 being the worst pain they can imagine. Results reported are an average of reported VAS scores for the 28 subjects who completed both phase I and phase II of the study.
Time Frame: 2 weeks
Population: Only subjects
Measure: Mean (Standard Deviation); unit: Visual Analog Scale
Groups:
- Placebo: All subjects who recieved Placebo lotion in either Phase I or II were considered.
Arm/Group | Pennsaid | Placebo
Number analyzed (Participants) | 28 | 28
Visual Analog Scale | 2.9 (2.6) | 4.3 (2.8)

3. Secondary Outcome: Clinical Neuropathic Pain Features- Constant Pain and Hypersensitivity After Treatment
Description: Subjects rated their "constant pain" and "hypersensitivity" using the Visual Analog Scale after a 2 week phase of using pennsaid lotion and after a 2 week phase of using placebo lotion.
  The Visual Analog Scale is subject reported on a scale of 0-10 with 0 being no pain, and 10 being the worst pain they can imagine. Results reported are an average of reported VAS scores for the 28 subjects who completed both phase I and phase II of the study.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Visual Analog Scale
Arm/Group | Pennsaid | Placebo
Number analyzed (Participants) | 28 | 28
Visual Analog Scale | 4.0 (2.9) | 4.3 (2.8)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the length of a subject's participation in the study (5 weeks).
Description: Due to the study design, subjects who withdrew before completing the entire study were not considered for any treatment period that they did not participate in due to drop out or withdrawl. Subjects who completed only part of a treatment period were considered.These numbers may differ from the total number enrolled in the study for this reason.
Groups:
- Pennsaid: Pennsaid (20-40 drops; 2-4 times daily for 2 weeks).
- Placebo: Placebo lotion (20-40 drops; 2-4 times daily for 2 weeks).
Arm/Group | Pennsaid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 0/32 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No